CLINICAL TRIAL: NCT04341233
Title: Enhanced Clinics for Patients Diagnosed With Ankylosing Spondylitis and Psoriatic Arthritis
Acronym: ECAP
Status: Withdrawn | Type: Observational
Why Stopped: withdrawn pre approvals
Sponsor: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: IRAS No: 265399
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Spondylitis, Ankylosing; Psoriatic Arthritis
Keywords: Nurse-Led Service; Enhanced Clinics
MeSH Terms: conditions — Spondylitis, Ankylosing; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The 19.5 months project will pilot the introduction of a hospital-based, nurse-led ankylosing spondylitis (AS) and psoriatic arthritis (PsA) service for patients being initiated on biologic therapy in NHS Lothian Edinburgh Western General Hospital.

It is anticipated that this new model of care will improve:

1. The time from referral for biologic therapy to initiation of treatment with a biological therapy due to the dedicated nurse to see patients
2. The management and monitoring of AS and PsA patients post commencement of treatment , in line with The National Institute for Health and Care Excellence (NICE) guidelines

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of AS or PsA
* Referral for initiation of biological therapy by patients regular consultant
* Age 18 years or older
* Willing and able to give informed consent

Exclusion Criteria:

· Unable to comply with study procedures

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of ankylosing spondylitis or psoriatic arthritis requiring initiation of biologic therapy.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2022-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Setup a nurse-led clinic | 3 months
  Appointing a nurse and training in biologic and DMARD counselling, clinical measures and clinic administration.
Develop and setup a tool, an NHS Lothian Excel database | 19.5 months
  Database enables trust to record data on the time taken to commence treatment with a biologic therapy from the point of initial referral to biologic therapy.
Develop and setup a tool, an NHS Lothian Excel database | 19.5 months
  Database enables trust to audit the results of the existing service for AS and PsA patients within the department (based on a cohort of 60 patients most recently initiated on biologics treatment within the department).
Develop and setup a tool, an NHS Lothian Excel database | 19.5 months
  Database enables trust to audit the results of the implementation of the clinic within the department.
Develop and setup a tool, an NHS Lothian Excel database | 19.5 months
  Database enables trust to assist with demonstrating that the care of patients within the clinic is in accordance with the NICE clinical guidelines and that there has been a reduction in the time to initiate biologic therapy at the end of the project against the baseline assessment.
Develop and setup a tool, an NHS Lothian Excel database | 19.5 months
  Database enables trust to develop a patient referral pathway into a new model of AS and PsA patient care, specifically in the nurse-led clinic.
Develop and setup a tool, an NHS Lothian Excel database | 19.5 months
  Database enables trust to utilise the new nurse-led clinic to improve consistency of care by reviewing and optimising biologic therapy for all new AS and PsA patients within the department according to NICE guideline recommendations.
Develop and setup a tool, an NHS Lothian Excel database | 19.5 months
  Database enables trust to use the evaluated model of care to enable NHS Lothian to build an informed business case to fund the continuation of this service in the future and expand it to all patients in their current service.

CONTACTS AND LOCATIONS:
Overall Officials: Neil McKay, Dr, Principal Investigator — NHS Lothian

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: National Institute for Health and Care Excellence (2016) Spondyloarthritis in over 16s: Diagnosis and management (NICE Guideline NG65). — https://www.nice.org.uk/guidance/ng65/chapter/recommendations